CLINICAL TRIAL: NCT05042856
Title: A Prospective, Single Center Study to Evaluate IOL Position, Clinical Outcome of PanOptix in High Myopic Cataract Patients
Brief Title: To Evaluate IOL Position, Clinical Outcome of PanOptix in High Myopic Cataract Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZYY-PanOptix IOL
Record Dates: First submitted 2021-08-22; First posted 2021-09-13 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Cataract; High Myopia
Keywords: PanOptix IOL; high myopic cataract patients
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PanOptix (Experimental): All the patients will be bilaterally implanted with PanOptix IOL，one eye will be randomized selected for monocular analysis of each patient.
  Interventions: Procedure: PanOptix IOL implantation

INTERVENTIONS:
Procedure: PanOptix IOL implantation — All the patients will be bilaterally implanted with PanOptix IOL，one eye will be randomized selected for monocular analysis of each patient.

SUMMARY:
To evaluate IOL position, clinical outcome of PanOptix in high myopic cataract patients

DETAILED DESCRIPTION:
A prospective, single center study to evaluate IOL position, clinical outcome of PanOptix in high myopic cataract patients.

The objective of this study to investigate the refractive and visual performance of PanOptix and explore their correlation with ELP change, capsular bending formation, IOL tilt/decentration in high myopic cataract patients.

PanOptix IOL provides good refractive outcomes and visual quality because of few ELP change, fast capsular bending formation and few tilt and decentration in high myopic cataract patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* 26 ≤Axial length<30mm, IOL power ≥6D (PanOptix IOL power is available +6D-+30D )
* Eyes with corneal astigmatism less than 1.0D (IOLMaster 700, Carl Zeiss Meditec AG)
* Eyes with pupil diameter between 3 and 5.5 mm (iTrace, Tracey Technology, Houston, Texas, USA)
* Eyes with angle kappa and angle Alpha ≤0.50 mm (iTrace);
* Eyes with corneal spherical aberration ≤ 0.50 (Pentacam).

Exclusion Criteria:

* Irregular corneal astigmatism
* Serious intraoperative complications, glaucoma, pseudoexfoliation syndrome, uveitis, macular degeneration or other retinal impairment
* Moderate-severe dry eye, corneal scarring, amblyopia
* Patients who can't cooperate with post-op 3 months follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Effective Lens Position（ELP） | 3 months
  Mean change of ELP for 3 months

SECONDARY OUTCOMES:
capsule bending index（CBI） | 3months
  Post-op 1 day，1week，1month，and 3 months monocular CBI(Swept source OCT,Casia SS-1000; Tomey)
lOL tilt | 3 months
  Post-op 1 day ,1 week,1 month and 3 months lOL tilt(Swept source OCT,Casia SS-1000; Tomey)
lOL decentration | 3 months
  Post-op 1 day ,1 week,1 month and 3 months lOL decentration(Swept source OCT,Casia SS-1000; Tomey)
Monocular uncorrected distance visual acuity（UDVA） | 3 months
  Pre-op and post-op 1 day,1 week,1 month and 3 months Monocular UDVA(Chinese standard logarithmic charts)
Monocular best corrected distance visual acuity（BCDVA）(5m) | 3 months
  Pre-op and post-op 1 day,1 week,1 month and 3 months Monocular BCDVA(5m)(Chinese standard logarithmic charts)
Monocular uncorrected intermediate visual acuity（UIVA） | 3 months
  Pre-op and post-op 1 day,1 week,1 month and 3 months Monocular UIVA(Chinese standard logarithmic charts)
Monocular distance corrected intermediate visual acuity(DCIVA)(60cm) | 3 months
  Pre-op and post-op 1 day,1 week,1 month and 3 months Monocular DCIVA(60cm)(Chinese standard logarithmic charts)
Monocular uncorrected near visual acuity（UNVA） | 3 months
  Pre-op and post-op 1 day,1 week,1 month and 3 months Monocular UNVA(Chinese standard logarithmic charts)
Monocular distance corrected near visual acuity(DCNVA)(40cm) | 3 months
  Pre-op and post-op 1 day,1 week,1 month and 3 months Monocular DCNVA(40cm)(Chinese standard logarithmic charts)
manifest refraction | 3 months
  Pre-op and post-op 1 day,1 week,1 month and 3 months manifest refraction
Monocular defocus curve | 3 months
  Post-op 1month,3 months monocular defocus curve
modulation transfer function（MTF） | 3 months
  Post-op 1 day,1 week,1 month and 3 months MTF(OPD-Scan III Analyzer,NIDEK CO.,LTD.,Tokyo,Japan)
high-order aberrations（HOA） | 3 months
  Post-op 1 day,1 week,1 month and 3 months HOA(OPD-Scan III Analyzer,NIDEK CO.,LTD.,Tokyo,Japan)

CONTACTS AND LOCATIONS:
Overall Officials: yune zhao, MD, Study Chair — Wenzhou Medical University
Locations (1):
- Ophthalmology and Optometry Hospital, Wenzhou, Zhejiang, China